CLINICAL TRIAL: NCT06572410
Title: Prospective Analysis of EnVisio Spatial Intelligence for Soft Tissue Localization and Guided Surgical Excision
Status: Recruiting | Type: Observational
Sponsor: Elucent Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 20242689
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Tumors, Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: Patient has selected breast conservation therapy
  Interventions: Device: EnVisio Navigation System

INTERVENTIONS:
Device: EnVisio Navigation System — Patient will be undergoing BCS Breast Conserving Surgery treatment for DCIS or invasive breast cancer with EnVisio Navigation System.

SUMMARY:
Observational study. The purpose of this study is to evaluate the use of real-time surgical navigation for the localization and surgical removal of soft tissue tumors. The goal is to collect information about the efficiency and effectiveness of the EnVisio Surgical Navigation for intraoperative guidance to obtain negative margin on initial specimen.

Prospective Patient Study: 200 consecutive patients

DETAILED DESCRIPTION:
Objectives

1.) To collect data throughout clinical patient workflow for evaluation of.

1. localization with SmartClip(s)
2. negative margin on primary specimen
3. specimen assessment
4. length of operation

The EnVisio® Navigation System was cleared as a Class II device by the FDA under 510(k) number K183400. The SmartClip® Soft Tissue Marker was cleared by the FDA under 510(k) number K180640.

Principal Investigator will receive monthly EnVisio system data from Company representative on the EnVisio system data collection for procedural cross reference resulting in.

* Date
* Time of SmartClip(s) auto detection
* Color and Number of SmartClip(s)
* Total time of EnVisio Guidance
* Specimen Assessment recordings of SmartClip to specimen edge as recorded by electrocautery tip on identified margin Medial/Lateral/Superior/Inferior/Anterior/Posterior)

Data will be collected from procedures performed including all imaging, clinical and pathologic outcomes. Pre and Post procedure data including number of individual lesions, localization of mass and number of SmartClips used. Patients planning surgical excision of an imaging identifiable in-breast will be offered entry into this study; the AdventHealth Winter Garden location will provide standard informed consent form for the purposes of this study. The projected accrual for this study is 200 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Patient has image identifiable lesion.
* Patient has selected breast conservation therapy IE: lumpectomy +/-radiation therapy, +/- chemotherapy +/- hormonal or targeted therapies. Neoadjuvant chemotherapy is not an exclusion criterion.
* Patient will be undergoing target tissue localization with the SmartClip
* Patient will be undergoing BCS Breast Conserving Surgery treatment for DCIS or invasive breast cancer with EnVisio ® Navigation System.
* Patient must be age > or = 18 years.
* Patients unable to provide consent to surgery must have authorized representative provide consent.

Exclusion Criteria:

* Patients undergoing mastectomy for resection of the targeted lesion.
* Patient is localized with an alternative method.
* Patient that are pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient will be undergoing BCS Breast Conserving Surgery treatment for DCIS or invasive breast cancer with EnVisio ® Navigation System
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Margin Positivity | Day of Surgery
  Specimen surgical resection volume gross measurements in 3 dimensions (length, width, depth) day of surgery.
  Definitive gross pathology results on final margin

CONTACTS AND LOCATIONS:
Locations (1):
- Advent Winter Garden, Winter Garden, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided